CLINICAL TRIAL: NCT05505097
Title: Open Randomized Comparative Crossover Study of the Safety and Pharmacokinetics of Dioxidin, Solution for Topical and External Use, 0.25 mg/ml and Dioxidin, Solution for Infusion and External Use, 5 mg/ml in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of Dioxidin, Solution for Topical and External Use, 0.25 mg/ml and Dioxidin, Solution for Infusion and External Use, 5 mg/ml in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DIO-01-04-2021
Record Dates: First submitted 2022-07-19; First posted 2022-08-17 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ABCD-sequence (Other): Hydroxymethylquinoxalindioxyde administration in a sequence A-B-C-D during the corresponding study periods 1, 2, 3, and 4
  Interventions: Drug: Hydroxymethylquinoxalindioxyde
- BCDA-sequence (Other): Hydroxymethylquinoxalindioxyde administration in a sequence B-C-D-A during the corresponding study periods 1, 2, 3, and 4
  Interventions: Drug: Hydroxymethylquinoxalindioxyde
- CDAB-sequence (Other): Hydroxymethylquinoxalindioxyde administration in a sequence C-D-A-B during the corresponding study periods 1, 2, 3, and 4
  Interventions: Drug: Hydroxymethylquinoxalindioxyde
- DABC-sequence (Other): Hydroxymethylquinoxalindioxyde administration in a sequence D-A-B-C during the corresponding study periods 1, 2, 3, and 4
  Interventions: Drug: Hydroxymethylquinoxalindioxyde

INTERVENTIONS:
Drug: Hydroxymethylquinoxalindioxyde — Dioxidin (Hydroxymethylquinoxalindioxyde), solution for topical and external use, 0.25 mg/ml, applied as:
  A - single rinsing of the oropharynx with 15.0 ml of the drug solution for at least 30 seconds B - single irrigation of the oropharynx by spraying the preparation 4 times with a spray nozzle C - irrigation of the skin on the back by spraying the preparation 4 times from a distance of 10 cm on 1% of the body surface using a spray nozzle and exposing the solution for 30 minutes or D - Dioxidin (Hydroxymethylquinoxalindioxyde), solution for infusion and external application, 5 mg/ml, single intravenous 5 mg/ml in 1 ml
  Other Names: Dioxidin

SUMMARY:
The study aimed for:

1. To study the safety of the drug Dioxidin, solution for topical and external use;
2. To determine the concentrations of the active substance of the studied drugs Dioxidin, solution for topical and external use, and Dioxidin, solution for infusion and external use in discrete time intervals;
3. To study pharmacokinetics of the drug Dioxidin, solution for topical and external application;
4. To determine the absolute bioavailability of the drug Dioxidine, solution for topical and external use.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary and handwritten informed consent form signed by a healthy volunteer to participate in the study before any of the study procedures
* Age from 18 to 45 years (inclusive)
* Verified diagnosis "healthy" by standard clinical, laboratory, instrumental methods of examination
* Blood pressure level: systolic from 100 to 130 mmHg, diastolic from 60 to 90 mmHg (inclusive)
* Heart rate 60 to 90 beats per minute (inclusive)
* Body mass index (BMI) is 18.5 ≤ BMI ≤ 30.0 kg/m², with a body weight of ≥55 kg for men and ≥45 kg for women
* Volunteers must behave appropriately, coherent speech must be observed
* For women of childbearing potential, negative pregnancy test; consent of volunteers to either abstain from sexual intercourse or use a dual barrier method of contraception for the duration of study participation, beginning with the Screening Period, and for 3 weeks after study termination
* Ability to follow the daily routine and dietary regimen of the study protocol
* Ability to attend all scheduled appointments and stay at the Research Center for all Study Periods

Exclusion Criteria:

* A history of allergic reactions
* A history of drug intolerance to the active and/or excipients in the study medications
* Inability to successfully perform oropharyngeal rinse test
* Any chronic illnesses
* History of gastrointestinal surgery (except appendectomy)
* Acute infectious diseases less than 4 weeks prior to screening
* Taking medications that significantly affect hemodynamics and medications that affect liver function (barbiturates, omeprazole, cimetidine, etc.) less than 2 months before screening
* Regularly taking medications less than 2 weeks before screening and taking a single medication 7 days before screening
* Donating blood (450 mL of blood or plasma or more) less than 3 months before screening
* For women, the last intake of oral contraceptives at least 2 months prior to screening
* Pregnant and lactating women, and women and men of childbearing age who cannot or do not abstain from sexual intercourse or use a dual barrier method of contraception for the duration of study participation, beginning with the Screening Period, and for 3 weeks after the study ends
* Participation in another clinical trial less than 3 months before screening or concurrently with this study
* Taking more than 10 units of alcohol (1 unit of alcohol is equivalent to 330 ml of beer, 150 ml of wine, or 40 ml of spirits) in the week in the last month before inclusion in the study or anamnestic evidence of alcoholism, drug abuse, or medication abuse
* Smoking more than 10 cigarettes per day currently, or a history of smoking this number of cigarettes in the 6 months prior to screening
* A positive blood test for HIV, syphilis, hepatitis B/C
* A positive urine test for narcotics and powerful drugs
* Positive breath alcohol test
* Positive COVID-19 test
* Scheduled inpatient hospitalization during the study for any reason other than hospitalization as required by this protocol
* Inability or inability to meet the requirements of the protocol, including for physical, mental or social reasons, in the opinion of the Researcher
* Work/study regimen that is likely to make it impossible for the volunteer to complete the study and/or comply with the schedule of procedures
* Other conditions that, in the opinion of the Researcher, prevent the inclusion of the volunteer in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | From 0 to 16 hours after each drug application on day 1, 7, 14, and 21 of the study
  Maximum plasma concentration (Cmax) of Hydroxymethylquinoxalindioxyde (HMQD)
Pharmacokinetics - tmax | From 0 to 16 hours after each drug application on day 1, 7, 14, and 21 of the study
  Time to reach Cmax (tmax) of HMQD
Pharmacokinetics - tlag | From 0 to 16 hours after each drug application on day 1, 7, 14, and 21 of the study
  Time from administration to first accessible concentration of HMQD
Pharmacokinetics - Vd | From 0 to 16 hours after each drug application on day 1, 7, 14, and 21 of the study
  Volume of distribution of HMQD
Pharmacokinetics - AUC0-t | From 0 to 16 hours after each drug application on day 1, 7, 14, and 21 of the study
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t) of HMQD
Pharmacokinetics - AUC0-inf | From 0 to 16 hours after each drug application on day 1, 7, 14, and 21 of the study
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) of HMQD
Pharmacokinetics - AUCextr | From 0 to 16 hours after each drug application on day 1, 7, 14, and 21 of the study
  Extrapolated AUC of HMQD, defined as (AUC0-inf - AUC0-t)/AUC0-inf
Pharmacokinetics - kel | From 0 to 16 hours after each drug application on day 1, 7, 14, and 21 of the study
  Elimination constant (kel) of HMQD
Pharmacokinetics - t1/2 | From 0 to 16 hours after each drug application on day 1, 7, 14, and 21 of the study
  Elimination half-life (t1/2) of HMQD
Pharmacokinetics - MRT | From 0 to 16 hours after each drug application on day 1, 7, 14, and 21 of the study
  Mean residence time (MRT) of HMQD

SECONDARY OUTCOMES:
Safety and Tolerability: adverse event (AE) rate | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to 43 days for each participant
  Number and frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: serious adverse event (AE) rate | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to 43 days for each participant
  Number and frequency of serious AEs (SAEs)
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | Screening, -10 h, -1 h, 2 h, 12, and 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | Screening, -10 h, -1 h, 2 h, 12, and 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  DBP, mmHg
Safety and Tolerability: vital signs - respiratory rate (RR) | Screening, -10 h, -1 h, 2 h, 12, and 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  RR, breaths per minute
Safety and Tolerability: vital signs - heart rate (HR) | Screening, -10 h, -1 h, 2 h, 12, and 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | Screening, -10 h, -1 h, 2 h, 12, and 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Body temperature, centigrade scale
Safety and Tolerability: physical examination results | Screening, -10 h, -1 h, 2 h, and 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Physical examination will follow the general rules of internal medicine: general examination, examination of mucous membranes and skin, including palpation of lymph nodes, evaluation of the musculoskeletal system, palpation, percussion, and auscultation of the main organ systems (cardiovascular, respiratory, digestive, and urinary systems) will be performed sequentially.
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screening and the end of the study or an early termination visit, whichever came first, within 43 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screening and the end of the study or an early termination visit, whichever came first, within 43 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: PQ interval (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screening and the end of the study or an early termination visit, whichever came first, within 43 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QRS complex (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval (QTc) | Screening and the end of the study or an early termination visit, whichever came first, within 43 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QTc (ms)
Safety and Tolerability: complete blood count - hemoglobin | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Hemoglobin, g/dL
Safety and Tolerability: complete blood count - red blood cells | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Red blood cells, 10^6/uL
Safety and Tolerability: complete blood count - hematocrit | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Hematocrit, %
Safety and Tolerability: complete blood count - platelets | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Platelets, 10^3/uL
Safety and Tolerability: complete blood count - white blood cells | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and at the end of the study or at early termination visit within the time frame of the study
  White blood cells, 10^3/uL
Safety and Tolerability: complete blood count - erythrocyte sedimentation rate | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Erythrocyte sedimentation rate, mm per hour
Safety and Tolerability: complete blood count - lymphocytes | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Lymphocytes, %
Safety and Tolerability: complete blood count - eosinophils | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Eosinophils, %
Safety and Tolerability: complete blood count - monocytes | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Monocytes, %
Safety and Tolerability: complete blood count - basophils | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Basophils, %
Safety and Tolerability: complete blood count - neutrophils | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Neutrophils, % (segmented and stab)
Safety and Tolerability: blood test results - glucose | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Glucose in blood serum, mmol/L
Safety and Tolerability: blood test results - total cholesterol | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Total cholesterol in blood serum, mmol/L
Safety and Tolerability: blood test results - total protein | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Total protein in blood serum, g/L
Safety and Tolerability: blood test results - total bilirubin | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Total bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - creatinine | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Creatinine in blood serum, umol/L
Safety and Tolerability: blood test results - alkaline phosphatase (ALP) | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  ALP in blood serum, U/L
Safety and Tolerability: blood test results - alanine transaminase (ALT) | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  ALT in blood serum, U/L
Safety and Tolerability: blood test results - aspartate transaminase (AST) | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  AST in blood serum, U/L
Safety and Tolerability: blood test results - aldosterone | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Aldosterone in blood serum, pmol/L
Safety and Tolerability: blood test results - cortisol | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and at the end of the study or at early termination visit within the time frame of the study
  Cortisol in blood serum, pmol/L
Safety and Tolerability: urinalysis - specific gravity | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Specific gravity of the urine
Safety and Tolerability: urinalysis - color | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Color of the urine
Safety and Tolerability: urinalysis - transparency | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Transparency of the urine
Safety and Tolerability: urinalysis - pH | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  pH of the urine
Safety and Tolerability: urinalysis - protein | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Protein in the urine (g/L)
Safety and Tolerability: urinalysis - glucose | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Glucose in the urine (mmol/L)
Safety and Tolerability: urinalysis (microscopy) - red blood cells | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Red blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - white blood cells | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  White blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - epithelial cells | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Epithelial cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - cylinders | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Cylinders in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - bacteria | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Bacteria in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - mucus | Screening, 24 h after each drug application on day 1, 7, 14, and 21 of the study, and on the end-of-study visit or on the early termination visit, whichever came first, within 43 days of study participation
  Presence of mucus in the urine

CONTACTS AND LOCATIONS:
Locations (1):
- Limited Liability Company "X7 Clinical Research", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided